CLINICAL TRIAL: NCT07053774
Title: Intranasal and Intravenous Oxytocin for Analgesia to Noxious Heat Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00134089; 40010559 (Other Grant/Funding Number: National Institute of Neurological Disorders and Stroke)
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-06

CONDITIONS: Pain, Acute
Keywords: healthy volunteers; pain control; oxytocin
MeSH Terms: conditions — Acute Pain; Agnosia | interventions — Oxytocin; Saline Solution; methylparaben; propylparaben; sodium phosphate; Citric Acid; Sorbitol; Glycerol

STUDY DESIGN:
Intervention Model Description: Each participant will receive an intravenous (IV) infusion of study drug and self-administer intranasal study drug. At study visit two some participants will receive IV saline (placebo) and oxytocin (48 IU) intranasally and some will receive IV oxytocin (20 IU) saline (placebo) intranasally. At visit three, participants will receive the opposite treatment sequence they received at visit 2. The order of study days will be randomized.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The Wake Forest University School of Medicine research pharmacy will prepare solutions and dispense them on the day of each study using a randomization stratified by sex that will be concealed until the end of the clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous (IV) oxytocin and intranasal (IN) placebo first (Experimental): On Visit 2 participants will receive IV infusion of oxytocin. At the beginning of the IV infusion, the participant will self-administer IN placebo.
  On Visit 3 participants will receive IV infusion of placebo. At the beginning of the IV infusion, the participant will self-administer IN oxytocin..
  Interventions: Drug: Intravenous oxytocin; Drug: Intravenous placebo; Drug: Intranasal oxytocin; Drug: Intranasal placebo
- Intravenous (IV) placebo and intranasal (IN) oxytocin first (Experimental): On Visit 2 participant will receive IV infusion of placebo. At the beginning of the IV infusion, the participants will self-administer IN oxytocin.
  On Visit 3 participants will receive IV infusion of oxytocin. At the beginning of the IV infusion, the participant will self-administer IN placebo.
  Interventions: Drug: Intravenous oxytocin; Drug: Intravenous placebo; Drug: Intranasal oxytocin; Drug: Intranasal placebo

INTERVENTIONS:
Drug: Intravenous oxytocin — Oxytocin, 10 International Units (IU) will be administered by IV infusion over 30 minutes and, 30 minutes later, a second 10 IU will be administered over 30 min, for a total dose of 20 IU. The first infusion will be at a rate of 0.125 IU/min for the first 5 min, then at 0.375 IU/min for the remaining 25 min. The second 30-min infusion will be at a fixed rate of 0.333 IU/min.
  Other Names: Pitocin
Drug: Intravenous placebo — Saline will be administered as two 30-min IV infusions separated by 30-min, using the same volume of infusion solution and rates of administration as in the intravenous oxytocin intervention.
  Other Names: Normal saline
Drug: Intranasal oxytocin — Oxytocin will be self-administered at the time the first IV infusion begins as a single 0.1 mL spray (12 IU) in each nostril followed in 5 min by another spray in each nostril. The total dose of oxytocin is 48 IU.
  Other Names: Pitocin
Drug: Intranasal placebo — Placebo (solution containing the excipients in the oxytocin solution but without oxytocin) will be self-administered at the time the first IV infusion begins as a single 0.1 mL spray in each nostril followed in 5 min by another spray in each nostril.
  Other Names: Excipients: chlorobutanol, methylparaben, propylparaben, dibasic sodium phosphate, anhydrous citric acid, sorbitol, glycerin, and sterile water

SUMMARY:
The goal of this research study is to find out how well oxytocin works to reduce pain. Oxytocin will be given intravenously (IV) and as a nasal spray. The study team also hopes to find out if the participants age, weight, or sex effects how well the study drug works.

Participants will be exposed to a heater on the skin at a training visit and rate how much pain different temperatures cause. On two separate visits, participants will use a nasal spray and get an IV infusion. After the IV and nasal spray, participants will rate the pain of the same skin heating temperature at various time points for 4 hours.

DETAILED DESCRIPTION:
This protocol will utilize a randomized, triple-masked, cross-over study design to compare intravenous (IV) to intranasal (IN) oxytocin administration for analgesia to an experimental pain stimulus in healthy volunteers. Equal numbers of adult men and women; ages 18-55 will be recruited. Participants will report to the research unit for three visits, 1) screening, informed consent, pregnancy test, and training to consistently rate pain from an FDA-approved device to test heat pain. The lowest temperature which causes a pain score of greater than 2 with 5 minutes of heating will be identified, 2) intravenous infusion and self-administered intranasal spray of study drug and 5-minute heat testing at intervals for 4 hours, 3) a repeat of the procedures done at visit two.

Participants will receive intravenous oxytocin, 20 IU and intranasal placebo on one of these visits and intravenous placebo and intranasal oxytocin, 48 IU, on the other. Pain score at the end of 5-minute skin heating will be compared using mathematical modeling of the time course of change in each individual and in the study population as a whole. The effect, if any, on these models of participant age, sex, and weight will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 and ≤75 years of age, Body Mass Index (BMI) <40.
* Generally in good health as determined by the Principal Investigator based on prior medical history, and as assessed to be American Society of Anesthesiologists physical status 1, 2, or 3.

Exclusion Criteria:

* Recent (<3 months) nasal surgery or chronic conditions requiring daily intranasal (IN) medications
* Hypersensitivity to any ingredient in Pitocin® (marketed preparation of oxytocin for parenteral injection)
* Latex allergy
* Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (e.g., active gynecologic disease in which increased tone would be detrimental such as uterine fibroids with ongoing bleeding)
* Women who are pregnant, are currently nursing or lactating, or have been pregnant within 2 years
* Neuropathy, chronic pain (located in any body location that is being treated), diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.
* Current or history of ventricular tachycardia, atrial fibrillation or prolonged QT interval.
* Past or current history of hyponatremia or at risk for hyponatremia; anyone taking thiazide diuretics, loop diuretics, combination diuretics, lithium, carbamazepine, enalapril, ramipril, celecoxib, temazepam, gliclazide, glimepiride, glibenclamide, glipizide, omeprazole, pantoprazole, desmopressin, serotonin selective reuptake inhibitors (SSRI's), monamine oxidase inhibitors (MAOI), or the recreational drug ecstasy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Pain Scale Score - End of 5-minute Skin Heating | Baseline Up to Hour 4.5
  Change in verbal pain scale score. Range is 0-10. 0 is equivalent to no pain and 10 is equivalent to the worst pain imaginable.
Pain Scale Score - During Skin Heating | Minute 5 During Skin Heating
  Verbal pain scale range is 0-10. 0 is equivalent to no pain and 10 is equivalent to the worst pain imaginable.

SECONDARY OUTCOMES:
Pain Scale Score - During Skin Heating | Minute 1 During Skin Heating
  Verbal pain scale range is 0-10. 0 is equivalent to no pain and 10 is equivalent to the worst pain imaginable.
Pain Scale Score - During Skin Heating | Minute 2 During Skin Heating
  Verbal pain scale range is 0-10. 0 is equivalent to no pain and 10 is equivalent to the worst pain imaginable.
Pain Scale Score - During Skin Heating | Minute 3 During Skin Heating
  Verbal pain scale range is 0-10. 0 is equivalent to no pain and 10 is equivalent to the worst pain imaginable.
Pain Scale Score - During Skin Heating | Minute 4 During Skin Heating
  Verbal pain scale range is 0-10. 0 is equivalent to no pain and 10 is equivalent to the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Atrium Health Wake Forest Baptist
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States